CLINICAL TRIAL: NCT04177524
Title: An Informatics Approach to Preventing Distracted Driving
Brief Title: Distracted Driving App Study for Teens and Parents/Caregivers
Acronym: IDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Minnesota HealthSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19-016717
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Distracted Driving

STUDY DESIGN:
Intervention Model Description: This study will utilize a crossover design with randomized assignment to three study arms to allow for comparison of app modes within drivers as each driver will act as their own control. The three app modes are: Background Mode (app runs in background and participants do not lock/unlock the phone), Manual Mode (participants manually unlock the phone), and Auto-Detect Mode (participants are automatically locked out of their phone if their phone camera detects them to be a driver or are automatically allowed to use their phone if the camera detects them to be a passenger).
Masking Description: Participants are aware of the differences between the app modes, and that the order in which they test out the different app modes is randomly assigned to them. The study team is not blinded to which study arm participants are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Participants alternate between using the Manual Mode of the app for 2 weeks and Auto-Detect Mode of the app for 2 weeks, for a total of 4 periods (8 weeks).
  Interventions: Device: Manual Mode; Device: Auto-Detect Mode
- Arm 2 (Experimental): Participants use the Auto-Detect Mode of the app for 4 weeks, followed by the Manual Mode for 4 weeks.
  Interventions: Device: Manual Mode; Device: Auto-Detect Mode
- Arm 3 (Experimental): Participants use the Background Mode of the app for 4 weeks, followed by the Auto-Detect Mode of the app for 4 weeks.
  Interventions: Device: Background Mode; Device: Auto-Detect Mode

INTERVENTIONS:
Device: Background Mode — The LifeSaver app tracks the date, time, and global positioning system (GPS) location of each trip that the participant takes in a moving vehicle, along with a list of apps used during the trip, but does not contain any anti-distracted driving features.
  Other Names: Mode 1
  Arms: Arm 3
Device: Manual Mode — In addition to the features in the Background Mode, the LifeSaver app locks the participants' phone while they are in a moving vehicle unless they actively press an "Emergency Unlock" or "Passenger Unlock" button.
  Other Names: Mode 2
  Arms: Arm 1; Arm 2
Device: Auto-Detect Mode — In addition to the features in Manual Mode, the LifeSaver app's "Passenger Unlock" feature can only be used if the app, via the smartphone's camera, confirms that the participant is not the driver of the vehicle.
  Other Names: Mode 3

SUMMARY:
The purpose of this research study is to determine if a new smartphone application helps to decrease distracted driving, and to learn about parent and teen perspectives about the application

DETAILED DESCRIPTION:
This 3-group randomized controlled trial aims to (1) evaluate the frequency of smartphone use among young drivers and their parents/caregivers while driving; and (2) determine if the LifeSaver mobile app reduces the rate of smartphone use while driving. Eligible participants will be licensed teenage drivers between the ages of 16 and 18 years, and a parent/caregiver. The app will be downloaded and installed on both parent/caregivers' and teens' phones to monitor phone use while in a vehicle for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Licensed teen drivers 16 years to 18 years and one parent/caregiver
* Teen and parent/caregiver are both Android smartphone users
* Teen and parent/caregiver both drive a minimum of 2 days per week

Exclusion Criteria:

* Non-fluency in written or spoken English

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Change in frequency of smartphone use while driving | Week 2, 4, 6, and post-intervention at Week 8
  Frequency of smartphone use is recorded by the LifeSaver app among the three app modes. Within-driver smartphone use over the 8-week study period is compared as the app modes change.

SECONDARY OUTCOMES:
Change in frequency of self-reported smartphone use while driving | Weeks 2, 4, 6, and Post-Intervention at Week 8
  The change in self-reported smartphone use while driving will be assessed using the same within-driver and between-driver comparisons as the primary outcome measure. Self-reported smartphone use is collected through 10 items on a participant survey that is completed at enrollment, Weeks 2, 4, 6 and post-intervention at Week 8. Participants report how many days during the previous 2 weeks (0-14) that they drove, and talked on a hands-held smartphone, talked on a hands-free smartphone, sent a text, and read a text while driving. Participants also report how many times per day (free text, any number greater than or equal to 0) that they drove, and talked on a hands-held smartphone, talked on a hands-free smartphone, sent a text, and read a text while driving. There is no overall self-reported smartphone use score for these survey items.
Participant acceptability of the smartphone App: survey | Post-Intervention at Week 8
  Participant assessment of accessibility will be collected, and Manual Mode and Auto-Detect Mode of the LifeSaver app will be compared. Participants complete a survey at Week 8, post-intervention. 8 items in the survey ask participants about accessibility of the app through Likert scales (range from Not at all to Extremely). 3 items in the survey ask participants about accessibility of the app through open-ended questions, where participants are able to enter free text. There is no overall score for these survey items.
Participant usability of the smartphone app: survey | Post-Intervention at Week 8
  Participant assessment of usability will be collected, and Manual Mode and Auto-Detect Mode of the LifeSaver app will be compared. Participants complete a survey at Week 8, post-intervention. 8 items in the survey ask participants about usability of the app through Likert scales (range from Not at all to Extremely). 3 items in the survey ask participants about usability of the app through open-ended questions, where participants are able to enter free text. There is no overall score for these survey items.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Curry, PhD, MPH, Principal Investigator — Children's Hospital of Philadelphia; Sara Seifert, MPH, Principal Investigator — Minnesota HealthSolutions
Locations (1):
- Children's Hospital of Philadelphia Roberts Center for Pediatric Research, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and study documents will be shared with Minnesota HealthSolutions (the sponsor). No identifiable data will be used for future studies without first obtaining CHOP Institutional Review Board (IRB) approval. The investigator will obtain a data use agreement between the provider (the PI) of the data and any recipient researchers (including others at CHOP) before sharing a limited dataset (PHI limited to dates and zip codes).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The study will comply with CHOP's data retention policy. All study data will be maintained for at least 6 years following study completion. There is no set timeline for the destruction of the study's de-identified data.
Access Criteria: IRB approval, data use agreement

DOCUMENTS (1):
  • Informed Consent Form (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT04177524/ICF_000.pdf